CLINICAL TRIAL: NCT04291586
Title: The Impact of Using an Interactive System and a Paper and Pencil Program in Psychosocial Rehabilitation of Psychiatric Patients
Brief Title: Comparing the Impact of Virtual Reality and Paper and Pencil on Psychosocial Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Irmãs Hospitaleiras Sagrado Coração de Jesus (Other)
Collaborators: Universidade da Madeira (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Casa de Saúde Câmara Pestana
Record Dates: First submitted 2019-05-24; First posted 2020-03-02 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Psychiatric Disease
Keywords: Virtual Reality; Cognitive Rehabilitation; Psychosocial Rehabilitation; Ecological validity; Personalization
MeSH Terms: conditions — Mental Disorders | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The Virtual Reality group will perform personalized activities of daily living in the context of a simulated city (Reh@City). The interaction with the virtual environment will be through a natural user interface.
  Interventions: Other: Virtual reality
- Paper and Pencil (Active Comparator): The paper and pencil group will perform a set of cognitive paper and pencil tasks personalized to their deficits and generated automatically through a Task Generator.
  Interventions: Other: Paper and Pencil

INTERVENTIONS:
Other: Virtual reality — Virtual Reality Intervention of 30 minutes, 3 times a week until reaching 24 sessions.
  Arms: Virtual Reality
Other: Paper and Pencil — Paper and Pencil Intervention of 30 minutes, 3 times a week until reaching 24 sessions.
  Arms: Paper and Pencil

SUMMARY:
Virtual Reality allows the integration of cognitive rehabilitation in a more ecologically valid context.

The purpose of this study is to determine whether this methodology has more impact on psychosocial rehabilitation than a paper and pencil personalized program.

DETAILED DESCRIPTION:
Cognitive impairments are frequently present on many psychiatric diseases, such as schizophrenia, depression, etc. and are not always given sufficient attention despite its limitations in activities of daily living (ADL's). Current cognitive rehabilitation methods mostly rely on paper-and-pencil tasks targeting isolated domains, which is not consistent with everyday life, and have limited ecological validity.

Virtual Reality (VR) has shown to be a solution for the development of accessible and ecologically valid systems but, does it have more impact than a paper and pencil personalized intervention?

Through a participatory design approach, with health professionals, the investigators have developed:

a motor-accessible and cognitive-personalized VR-based system, where conventional cognitive tasks were operationalized in meaningful simulations of ADL's (Reh@City) and; a web tool which generates personalized paper and pencil tasks (Task Generator).

The investigators goal is to have a sample of 30 inpatients from a psychosocial rehabilitation unit, with no age limit, randomly allocated in two groups: 1) the experimental group, where participants will perform 30 minutes of the VR training with Reh@City; and 2) the control group, where participants will perform 30 minutes of the paper and pencil training with the Task Generator.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients of psychosocial rehabilitation unit;
* Cognitive deficit but with enough capacity to understand the task and follow instructions;
* Able to read and write.

Exclusion Criteria:

* Patients experiencing an acute psychiatric episode.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (Cognitive Screening) | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Montreal Cognitive Assessment. Higher values represent better outcomes.

SECONDARY OUTCOMES:
Toulouse-Pieron (Attention) | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Toulouse-Pieron Cancellation Test.
Semantic Fluency and Phonemic Fluency Tests | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Semantic Fluency and Phonemic Fluency Tests
Verbal Paired Associates (WMS-III) (Memory) | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Verbal Paired Associates (WMS-III)
Rey Complex Figure | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Rey Complex Figure
Symbol Search and Coding (WAIS III) | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Symbol Search and Coding (WAIS III)
Rey 15-Item Memory Test | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Rey 15-Item Memory Test

OTHER OUTCOMES:
Beck Depression Inventory - II | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Beck Depression Inventory - II. It is a self-report inventory that aims to measure the severity of depression. Can be scored between 0-63. Minimal depression, 0-11; Mild depression, 12-18; Moderate depression, 19-24; Severe depression, above 25.
Barthel Index | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Barthel Index. It's a scale that measures functionality, with features of activities of daily living with the item: bowel control, bladder control, personal hygiene, using the toilet, eating, transferring, walking on a level surface, getting dressed and undressed, going up and down stairs, taking a shower. The maximum score obtainable is 100 points: scores between 91-99, correspond to slight dependence; 61-90, to moderate dependence; 21-60, to serious dependence; and 0-20, to total dependence.
Katz Index | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the Katz Index. It's a scale that measures functionality, with features of activities of daily living with the item: showering, dressing, using the toilet, sphincter control, mobility and eating. The highest score obtainable is 6, corresponding to independent; scores between 3 and 5, correspond to moderate dependence; and scores below 2, correspond to very dependent.
World Health Organization Quality of Life - Bref (WHOQOL-Bref) - Quality of Life Assessment | Baseline, End (8 weeks) and 8-weeks follow-up
  Change from baseline in the WHOQOL-Bref Quality of Life Assessment. This scale is divided in four domains, physical health, social, psychological and environmental. For the physical health we use the questions: 3 (inverse), 4 (inverse),10,15, 16, 17, 18. For the psychological, questions: 5, 6, 7, 11, 19, 26 (inverse). For the social domain, the questions: 20, 21, 22. For the environmental domain, the questions: 8, 9, 12, 13, 14, 23, 24, 25. The main score is obtained through the sum of the four domains and higher scores correspond to higher perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sergi Bermudez, Ph,D, Principal Investigator — Madeira Interactive Technologies Institute
Locations (1):
- Instituto das Irmãs Hospitaleiras do Sagrado Coração de Jesus - Casa de Saúde Câmara Pestana, Funchal, Funchal-Madeira, Portugal

IPD SHARING:
Plan to Share IPD: No